CLINICAL TRIAL: NCT05853991
Title: Effects of Affective Touch, Therapeutic Touch (OMT), and Static/Nonspecific Touch on Brain Connectivity and Metabolic Biomarkers in Preterm Infants
Brief Title: Effects of Touch on Brain Connectivity and Metabolic Biomarkers in Preterm Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Come Collaboration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COME-23-01
Record Dates: First submitted 2023-02-07; First posted 2023-05-11 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Preterm; Infant ALL; Premature; Disease
MeSH Terms: conditions — Premature Birth; Disease | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic touch (Experimental): The intervention will be based on 2 phases: 1) assessment to identify areas following the NAME procedure, 2) treatment to improve the function of the area identified
  Interventions: Other: osteopathic manipulative treatment
- Affective touch (Active Comparator): Participants will receive an affective touch intervention following the standardised procedure for affective touch
  Interventions: Other: Active comparator
- Static touch (Placebo Comparator): Participants will receive a static touch intervention following the standardised procedure for static touch
  Interventions: Other: Placebo

INTERVENTIONS:
Other: osteopathic manipulative treatment — The intervention will be based on the specific assessment and treatment of the preterm developed by the team and validated through different studies.
  Arms: Therapeutic touch
Other: Active comparator — Application of affective touch
  Arms: Affective touch
Other: Placebo — Application of static touch
  Arms: Static touch

SUMMARY:
Improving the quality of life of preterm children by 2035 is the top priority of worldwide health organisations, including the WHO. Every year, 15 million preterm infants, particularly those under 32 weeks of age, are at significant risk of neurocognitive impairments with adverse health consequences (disability, developmental delay, disease), exacerbated by the lack of post-hospital care for newborns.

Intervening on the health of the preterm newborn through certain types of "touch" from its first days of life to activate its cutaneous senses permits, in reality, a significant improvement in the clinical state of the infant, hence promoting its growth, development, and social behaviour.

In the neonatal period, during which significant neurological development occurs, tactile interactions and close physical proximity between infants and caregivers have significant short-term effects on the health of premature infants (weight gain, brain and vision development) and medium- to long-term effects on their development and expression of sociability.

The likelihood that a premature newborn may develop attention and autism spectrum disorders, brain, gastrointestinal, and respiratory difficulties, as well as sleep disorders during the preschool years, is so high that clinical and social settings must prioritise care.

Utilizing functional magnetic resonance imaging (fRMI), computerized electroencephalogram (EEG), and metabolomics, the research aims to explore the effects of touch, including physiotherapy and manual therapy (OMT) approaches, on brain activity.

This research intends to examine the impact of touch on premature infants' brain activity (physical biomarker) and metabolic activity (biological biomarker).

ELIGIBILITY:
Inclusion Criteria:

* Preterm birth, between 32.0 and 33.6 weeks gestational age (GA);
* Absence of comorbidities that could affect the stability of vital parameters, and therefore represent a contraindication to the proposed intervention. Comorbities include sepsis, pathologies pertaining to surgery, respiratory or cardiovascular instability, birth from a drug-addicted or HIV-positive mother) or known congenital pathologies;
* Obtaining informed consent for participation in this research project from parents or legal guardians.

Exclusion Criteria:

* Preterm infants born before 32.0 weeks of GA and after 34 weeks and with respiratory and neurological pathologies and any additional comorbities.
* Children whose parents will not read and sign or in case of failure to obtain informed consent will be excluded from the study.

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
brain changes | 1 hour
  pre-post changes in BOLD levels among different brain areas

SECONDARY OUTCOMES:
electroencephalogram (EEG) changes | 10 days
  pre-post changes from baseline in the EEG power in slow delta waves band at the end of the treatment period
Proton Nuclear Magnetic Resonance Spectroscopy (1H NMR) at T1 | 1 hour
  pre-post changes in urinary metabolites as assessed by 1H NMR at T1
Proton Nuclear Magnetic Resonance Spectroscopy (1H NMR) at T2 | 4 days
  pre-post changes in urinary metabolites as assessed by 1H NMR at T2
Proton Nuclear Magnetic Resonance Spectroscopy (1H NMR) at T3 | 8 days
  pre-post changes in urinary metabolites as assessed by 1H NMR at T3
Proton Nuclear Magnetic Resonance Spectroscopy (1H NMR) at T4 | 12 days
  pre-post changes in urinary metabolites as assessed by 1H NMR at T4
Proton Nuclear Magnetic Resonance Spectroscopy (1H NMR) at T5 | 40 weeks
  pre-post changes in urinary metabolites as assessed by 1H NMR at T5
Mass Spectrometry combined with Liquid Chromatography (CL-MS)at T1 | 1 hour
  pre-post changes in urinary metabolites as assessed by CL-MS at T1
Mass Spectrometry combined with Liquid Chromatography (CL-MS)at T2 | 4 days
  pre-post changes in urinary metabolites as assessed by CL-MS at T2
Mass Spectrometry combined with Liquid Chromatography (CL-MS)at T3 | 8 days
  pre-post changes in urinary metabolites as assessed by CL-MS at T3
Mass Spectrometry combined with Liquid Chromatography (CL-MS)at T4 | 12 days
  pre-post changes in urinary metabolites as assessed by CL-MS at T4
Mass Spectrometry combined with Liquid Chromatography (CL-MS)at T5 | 40 weeks
  pre-post changes in urinary metabolites as assessed by CL-MS at T5
Mass Spectrometry combined with Gas Chromatography (CG-MS) at T1 | 1 hour
  pre-post changes in urinary metabolites as assessed by CG-MS at T1
Mass Spectrometry combined with Gas Chromatography (CG-MS) at T2 | 4 days
  pre-post changes in urinary metabolites as assessed by CG-MS at T2
Mass Spectrometry combined with Gas Chromatography (CG-MS) at T3 | 8 days
  pre-post changes in urinary metabolites as assessed by CG-MS at T3
Mass Spectrometry combined with Gas Chromatography (CG-MS) at T4 | 12 days
  pre-post changes in urinary metabolites as assessed by CG-MS at T4
Mass Spectrometry combined with Gas Chromatography (CG-MS) at T5 | 40 weeks
  pre-post changes in urinary metabolites as assessed by CG-MS at T5

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale dei bambini "Vittore Buzzi", Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manzotti A, Cerritelli F, Lombardi E, Tansini L, Pisanu D, Di Leo D, Vergani E, Righini A, Arrigoni F, Fanos V, Rescigno M, Veggiotti P, Lista G, Gazzolo D. Impact of touch interventions on brain activity in moderately preterm infants: study protocol for a pilot randomised controlled trial. BMJ Open. 2025 Oct 27;15(10):e102964. doi: 10.1136/bmjopen-2025-102964. PMID 41145247